CLINICAL TRIAL: NCT03316105
Title: Effect of T6 Dermatome Electrical Stimulation on Gastroduodenal Motility in Healthy Volunteers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Electrical device malfunction; recruitment was stopped.
Sponsor: Mayo Clinic (Other)
Collaborators: Elira Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-004101
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Results first posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transcutaneous electrical nerve stimulation (TENS) stimulation (Active Comparator): During this TENS unit stimulation arm, subjects will have a narrow tube (about the diameter of a telephone cord) placed into the subjects small intestine by the study physician and trained technician. The technician will use a small amount of fluoroscopy (radiation) to make sure the tube is placed in the proper position. About one hour after the tube has been placed subjects will be given a breakfast meal. The narrow tube (GDM) will take pressure readings after being placed. After four hours, subjects will again be given a second meal. Fifteen minutes of electrical stimulation will be given to subjects fifteen minutes before ingestion of lunch. After ingestion of lunch, 60 minutes of the electrical stimulation will be applied. When the test is done, the tube will be removed.
  Interventions: Device: Elira Investigational TENS device
- No TENS stimulation (Sham Comparator): During this no TENS unit stimulation arm, subjects will have a narrow tube (about the diameter of a telephone cord) placed into the subjects small intestine by the study physician and trained technician. The technician will use a small amount of fluoroscopy (radiation) to make sure the tube is placed in the proper position. About one hour after the tube has been placed subjects will be given a breakfast meal. The narrow tube (GDM) will record stomach pressure readings after being placed. After four hours, subjects will again be given a second meal. The TENS unit stimulation will be placed but no electrical stimulation will be given. When the test is done, the tube will be removed.
  Interventions: Device: Elira Investigational TENS device

INTERVENTIONS:
Device: Elira Investigational TENS device — TENS unit placed on skin will deliver electric stimulation to abdominal area.
  Other Names: Electric Stimulation from TENS unit

SUMMARY:
The investigators are doing this research study to find out the effect of T6 Dermatomal Electrical Stimulation (delivered by a Transcutaneous Electrical Nerve Stimulation (TENS) unit) on stomach motor activity.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers with BMI ≤34.99 kg/m^2 residing within 125 miles of Mayo Clinic in Rochester, Minnesota; these will be healthy individuals with no unstable psychiatric disease and not currently on treatment for cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, or endocrine (other than hyperglycemia on diet) disorders.
2. Women of childbearing potential will be using an effective form of contraception, and have negative pregnancy tests within 48 hours of the test day.
3. Subjects must have the ability to provide informed consent before any trial-related activities.
4. Eligible individuals will be asked to avoid taking additional medications and supplements for one week before and after the test day, unless reviewed and approved by the study team.

Exclusion Criteria:

1. Abdominal surgery other than appendectomy, Caesarian section or tubal ligation.
2. Positive history of chronic gastrointestinal diseases, systemic disease that could affect gastrointestinal motility, or use of medications that may alter gastrointestinal motility.
3. Positive history of spinal cord injury and/or chronic back pain.
4. Significant untreated psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Inventory (HAD). If such a dysfunction is identified by a HAD score >11 on either Anxiety or Depression or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up.
5. Intake of medication, whether prescribed or over the counter (except multivitamins), within 7 days of the study. Exceptions are birth control pill, estrogen replacement therapy, thyroxine replacement therapy, low dose analgesia or anti-inflammatory medications (Acetaminophen and Ibuprofen) and any medication administered for co-morbidities as long as they do not alter gastrointestinal motility.
6. Subjects may also be excluded from participation for other factors at the discretion of the principal investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, M.D, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcutaneous Electrical Nerve Stimulation (TENS) Stimulation | No TENS Stimulation
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TENS Unit Stimulation: During this TENS unit stimulation arm, subjects will have a narrow tube (about the diameter of a telephone cord) placed into the subjects small intestine by the study physician and trained technician. The technician will use a small amount of fluoroscopy (radiation) to make sure the tube is placed in the proper position. About one hour after the tube has been placed subjects will be given a breakfast meal. The narrow tube (GDM) will take pressure readings after being placed. After four hours, subjects will again be given a second meal. Fifteen minutes of electrical stimulation will be given to subjects fifteen minutes before ingestion of lunch. After ingestion of lunch, 60 minutes of the electrical stimulation will be applied. When the test is done, the tube will be removed.
  Elira Investigational TENS device: TENS unit placed on skin will deliver electric stimulation to abdominal area.
- No TENS Unit Stimulation: During this no TENS unit stimulation arm, subjects will have a narrow tube (about the diameter of a telephone cord) placed into the subjects small intestine by the study physician and trained technician. The technician will use a small amount of fluoroscopy (radiation) to make sure the tube is placed in the proper position. About one hour after the tube has been placed subjects will be given a breakfast meal. The narrow tube (GDM) will record stomach pressure readings after being placed. After four hours, subjects will again be given a second meal. The TENS unit stimulation will be placed but no electrical stimulation will be given. When the test is done, the tube will be removed.
  Elira Investigational TENS device: TENS unit placed on skin will deliver electric stimulation to abdominal area.
- Total: Total of all reporting groups
Arm/Group | TENS Unit Stimulation | No TENS Unit Stimulation | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (11.6) | 34 (7.9) | 36.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Effect of T6 Dermatomal Electrical Stimulation on Subjects Stomach Motor Activity
Description: Testing to see if dermatomal electrical stimulation will speed up or slow down the stomach motor activity.
Time Frame: through study completion, an average of 1 year
Population: Electrical device malfunction; recruitment was stopped.
Arm/Group | TENS Unit Stimulation | No TENS Unit Stimulation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed through study completion, an average of 1 year
Arm/Group | TENS Unit Stimulation | No TENS Unit Stimulation
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT03316105/Prot_SAP_000.pdf